CLINICAL TRIAL: NCT05200247
Title: Multi-centre, Open-label, Expanded Access Trial of Spesolimab i.v. in Patients With Generalized Pustular Psoriasis (GPP) Presenting With a Flare
Brief Title: An Expanded Access Trial in Japan to Provide Spesolimab to People With a Flare-up in Generalized Pustular Psoriasis Who Have no Other Treatment Options
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0073
Record Dates: First submitted 2022-01-11; First posted 2022-01-20 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spesolimab (Experimental)
  Interventions: Drug: spesolimab

INTERVENTIONS:
Drug: spesolimab — solution for infusion

SUMMARY:
This Expanded Access trial in Japan is open to people with a serious skin disease called Generalized Pustular Psoriasis (GPP). This program provides a medicine called spesolimab to people with a GPP flare-up who have no alternative treatment options.

Participants get a single infusion of spesolimab into a vein. They can get another spesolimab infusion one week after the first infusion if the doctors think it is helpful.

Participants are in the program for about 4 months and visit the study site about 5 to 6 times. The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of GPP confirmed based on the Japanese Dermatological Association (JDA) guidelines for the management and treatment of GPP.
* Patient is experiencing a flare, defined as new or worsening of widespread eruption of sterile macroscopically visible pustules, with or without systemic inflammation, as assessed by the investigator.
* Male or female patients, aged 18 to 75 years at time of enrollment. Women of childbearing potential (WOCBP) must be willing and able to use a highly effective method of birth control per International Council for Harmonization (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with International Council for Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* No satisfactory authorised alternative therapy exists, as assessed by the investigator.

Exclusion criteria

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

  -- Women who stop nursing before study drug administration do not need to be excluded from participating; they should refrain from breastfeeding for 16 weeks after the last spesolimab infusion.
* Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold Upper Level of Normal (ULN) elevation in Aspartate Transaminase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin.
* Active systemic infections (fungal and bacterial disease) during the last 2 weeks prior to drug administration, as assessed by the investigator.
* Increased risk of infectious complications (e.g. recent pyogenic infection, any congenital or acquired immunodeficiency (e.g. Human Immunodeficiency Virus (HIV)), past organ or stem cell transplantation), as assessed by the investigator.
* Relevant chronic or acute infections, including active tuberculosis (TB), HIV infection or viral hepatitis at the time of drug administration.

  * Patients should be evaluated for TB infection prior to initiating treatment with spesolimab.
  * Anti-TB therapy should be considered, in accordance with local guidelines, prior to initiating spesolimab in patients with latent TB or a history of TB.
* History of allergy / hypersensitivity to systemically administered spesolimab or its excipients.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Immediate life-threatening flare of GPP requiring intensive care treatment according to the investigator's judgement. Life-threatening complications include cardiovascular / cytokine driven shock, pulmonary distress syndrome, or renal failure.

Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Nagoya City University Hospital, Aichi, Nagoya
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Mie University Hospital, Mie, Tsu
  - Tohoku University Hospital, Miyagi, Sendai
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Teikyo University Hospital, Tokyo, Itabashi-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multicentre, single-arm trial designed to provide early access to spesolimab, for patients with generalised pustular psoriasis (GPP) presenting with a flare and for whom no satisfactory authorised alternative therapy existed and who were unable to participate in a clinical trial, as assessed by the investigator.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Spesolimab 900 mg i.v. SD: Patient with GPP flare received intravenously (i.v.) a single dose (SD) of 900 milligram (mg) of spesolimab on Day 1 of Week 1. A second dose of 900 mg spesolimab was administered one week after the initial infusion if deemed necessary by the investigator.
Period: Overall Study
Arm/Group | Spesolimab 900 mg i.v. SD
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: This patient set included all patients who received at least one dose of study drug.
Arm/Group | Spesolimab 900 mg i.v. SD
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: Number of patients with any treatment emergent adverse events (TEAEs) is reported.
  An adverse events (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.
  An AE that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
Time Frame: From first administration of study drug until last administration of study drug + 16 weeks of follow up, up to 6.3 months.
Population: Treated Set (TS): This patient set includes all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab 900 mg i.v. SD
Number analyzed (Participants) | 11
Participants | 7

2. Secondary Outcome: Occurrence of Treatment Emergent Serious Adverse Events (SAEs)
Description: Number of patients with treatment emergent serious adverse events (SAEs) is reported.
  A serious adverse event (SAE) was defined as any AE which fulfils at least one of the following criteria:
  * results in death,
  * is life-threatening, which refers to an event in which the patient was at risk of death at the time of the event;
  * requires inpatient hospitalisation or prolongation of existing hospitalisation,
  * results in persistent or significant disability or incapacity,
  * is a congenital anomaly / birth defect,
  * is deemed serious for any other reason if it is an important medical event when based on appropriate medical judgement which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.
  * An event that possibly leads to disability will be handled as 'deemed serious for any other reason' and, therefore, reported as an SAE.
Time Frame: as for outcome 1
Population: Treated Set (TS): This patient set includes all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab 900 mg i.v. SD
Number analyzed (Participants) | 11
Participants | 0

3. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events of Special Interest (AESIs)
Description: Number of patients with treatment emergent adverse events of special interest (AESIs) is reported.
  The term adverse events of special interest (AESI) relates to any specific adverse event (AE) that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class.
  The following are considered as AESIs:
  * Potential Severe Drug Induced Liver Injury (DILI)
  * Systemic hypersensitivity reactions including infusion reactions and anaphylactic reaction
  * Severe infections (according to RCTC grading in the ISF)
  * Opportunistic and mycobacterium tuberculosis infections
  * Peripheral neuropathy.
Time Frame: as for outcome 1
Population: Treated Set (TS): This patient set includes all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab 900 mg i.v. SD
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: From first administration of study drug until last administration of study drug + 16 weeks of follow up, up to 6.3 months.
Description: Treated Set (TS): This patient set includes all patients who received at least one dose of study drug.
Arm/Group | Spesolimab 900 mg i.v. SD
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab 900 mg i.v. SD (N=11)
Constipation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Face oedema (General disorders) | 1
Malaise (General disorders) | 1
Periodontitis (Infections and infestations) | 1
Wound (Injury, poisoning and procedural complications) | 1
Coronavirus test positive (Investigations) | 1
Transaminases increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT05200247/Prot_SAP_000.pdf